CLINICAL TRIAL: NCT06325865
Title: Perception of Unpleasant Sensations in Patients With Amyotrophic Lateral Sclerosis During Procedures Performed in Clinical Trials
Brief Title: Perception of Unpleasant Sensations During Study Procedures in ALS Patients
Acronym: PESALS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 23C305
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Study procedures
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Interview with ALS patient in which the experiences of unpleasant sensations or pain during study procedures are assessed in a qualitative manner.

SUMMARY:
Diagnosis of Amyotrophic Lateral Sclerosis (ALS) is considered a traumatic life event for both the patient and their next-of-kin/carers, due to the lack of treatment. Clinical Trials can offer pioneering treatment to reduce the impact of the disease and improve future treatments worldwide. Research protocols may involve routine diagnostic and/or therapeutic procedures which the patients may be already aware of and, therefore, expecting specific sensations. These could compromise participation or drop-out rate. Despite everything, participation in a clinical trial can guarantee continuity of care also thanks to the execution of these same procedures, through preferential access compared to other patients.

Aim of this study is to investigate the unpleasant sensations perceived by ALS patients during procedures in clinical trials. Analysing what type of pain/discomfort frightens patients during diagnostic and/or therapeutic procedures, including the different methods of administration of the study drug. Provide data to implement effective therapy and offer constant patients support throughout ALS specific and needed procedures. Evaluate if this support could influence adherence rate of ALS patients to conduct clinical trials as required. Provide information for future studies to create an ALS Clinical Trials multiple-retention-factors adherence scale. Create and implement an ALS-specific pain scale accounting for its impact on daily activities, aiding an interdisciplinary approach of pain management. Identify the best pain management strategies and compliance techniques to address ALS, not merely in clinical trials. Provide the best individualized care for ALS patients improving their quality of life and mental state.

This is a descriptive phenomenological study and data will be analyzed according to Sundler's method. Based on the experience of the researchers and the recommendations proposed by Sandelowski, a total of 20 interviews are estimated in order to reach the theoretical saturation per category of reference. Data collection will be carried out through in-depth semi-structured interviews recorded (13 open-ended questions after the execution of the procedures).

ELIGIBILITY:
Inclusion Criteria:

* Spinal or bulbar Amyotrophic Lateral Sclerosis (ALS)
* Age > 18 years
* Adequate understanding of Italian language
* Full understanding of the study
* Informed consent signed
* Current or past participation in interventional clinical studies
* Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) score of item # 4 ≥ 2, or score of item #1 ≥ 1

Exclusion Criteria:

* Clinically relevant cognitive dysfunction
* Inability to answer orally or by writing to the questions of the interview
* Hospital Anxiety and Depression Scale (HADS) scale ≥ 11

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Amyotrophic Lateral Sclerosis (ALS) patients who are currently participating in interventional clinical studies or who have particpated in the recent past.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Prevalence of experience of unpleasant sensations or pain | At enrollment
  Prevalence of reported experience of unpleasant sensations orn pain during study procedures
Study procedure that causes unpleasant sensations or pain | At enrollment
  Qualitative description of study procedure that causes unpleasant sensations or pain
Duration of unpleasant sensations or pain caused by the study procedure | At enrollment
  Duration in minutes of unpleasant sensations or pain caused by the study procedure

SECONDARY OUTCOMES:
HADS score | At enrollment
  Score on Hospital Anxiety and Depression Scale (HADS) scale
ALSFRS score | At enrollment
  Score on Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) scale

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico italiano IRCSS, San Luca Hospital, Milan, Italy